CLINICAL TRIAL: NCT01680835
Title: The US StuDy for EvalUating EndovasculaR TreAtments of Lesions in the Superficial Femoral Artery and Proximal Popliteal By usIng the EverfLex NitInol STent System Post Approval Study
Brief Title: EverFlex Post Approval Study
Acronym: DURABILITY PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-1001
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Peripheral Arterial Disease; Lower Extremity Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study cohort (Experimental): All patients enrolled in this study will be treated with the EverFlex™ Self-Expanding Peripheral Stent System.
  Interventions: Device: EverFlex™ Self-Expanding Peripheral Stent System

INTERVENTIONS:
Device: EverFlex™ Self-Expanding Peripheral Stent System — Using the EverFlex™ Self-Expanding Peripheral Stent System to treat atherosclerotic superficial femoral artery (SFA) and proximal popliteal lesions 4-18 cm long in subjects with Rutherford Clinical Categories 2-4.

SUMMARY:
This post-approval study is designed to confirm the long-term safety and effectiveness of the EverFlex™ Self-Expanding Stent System for the treatment of atherosclerotic superficial femoral artery (SFA) and proximal popliteal arteries.

ELIGIBILITY:
General Inclusion Criteria

1. Has stenotic, restenotic (from PTA or adjunct therapy, not including stents or stent grafts), or occluded lesion(s) located in the native superficial femoral artery or superficial femoral and proximal popliteal arteries suitable for primary stenting.
2. Has a Rutherford Clinical Category Score of 2, 3 or 4.
3. Is willing to comply with all follow-up evaluations at the specified times.
4. Is ≥ to18 years old.
5. Provides written informed consent prior to enrollment in the study.

Angiographic Inclusion Criteria Subjects must meet all of the following angiographic inclusion criteria. The implanting physician bases all angiographic inclusion criteria on visual determination at the time of the procedure.

1. Target lesion(s) located within the native SFA/proximal popliteal: distal point at least 3 cm above the cortical margin of the femur and proximal point at least 1 cm below the origin of the profunda femoralis measured by straight posteroanterior (PA) view for distal lesions, ipsilateral oblique view for proximal lesions.
2. Evidence of ≥ 50% stenosis or restenosis (from PTA or adjunct therapy, not including stents or stent grafts), or occlusion of target lesion(s).
3. Target lesion(s) total length is ≥ 4 cm and ≤ 18 cm.
4. Target vessel diameter is ≥ 4.5 mm and ≤ 7.5 mm.
5. There is evidence of at least one runoff vessel to the ankle/foot of the limb to be treated that does not also require treatment for significant (> 50% stenosis or occlusion) stenosis during the index procedure.

General Exclusion Criteria

1. Has undergone previous implantation of stent(s) or stent graft(s) in the target vessel.
2. Has a contraindication or known allergy to antiplatelet therapy, anticoagulants, thrombolytic drugs, contrast media or any other drug used in study according to the protocol.
3. Has known hypersensitivity to nickel-titanium.
4. Has bleeding diathesis, coagulopathy, known hypercoagulable condition, or refuses blood transfusion.
5. Female currently breastfeeding, pregnant, or of childbearing potential not using adequate contraceptive measures.
6. Has life expectancy of less than 1 year.
7. Has planned use of thrombectomy, atherectomy, brachytherapy or laser devices during procedure.
8. Has previously been enrolled in the DURABILITY PAS study.
9. Has received endovascular treatment of target lesion by percutaneous transluminal angioplasty or any other means of previous endovascular treatment (e.g. cutting balloon, scoring balloon, cryoplasty, thrombectomy, atherectomy, brachytherapy or laser devices) within six months of the index procedure.
10. Has any planned surgical intervention or endovascular procedure 14 days before or 30 days after the index procedure.
11. Is currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints.
12. Has any co-morbid condition that precludes endovascular treatment.

Angiographic Exclusion Criteria The subject must not meet any of the following angiographic exclusion criteria. The implanting physician bases all angiographic exclusion criteria on visual determination at the time of the procedure.

1. Exchangeable guidewire cannot cross the target lesion and/or re-enter true vessel lumen distal to lesion(s).
2. Presence of significant (> 50% stenosis or occlusion) ipsilateral common femoral stenosis.
3. Aneurysmal target vessel.
4. Presence of an acute intraluminal thrombus at the proposed lesion site.
5. Perforation, dissection or other injury of the access or target vessel requiring additional stenting or surgical intervention prior to start of PTA procedure.
6. Focal popliteal disease in the absence of femoral disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon S Matsumura, MD, Principal Investigator — University of Wisconsin, Madison; Krishna Rocha-Singh, MD, Principal Investigator — Prairie Heart Institute
Locations (23):
- United States (23):
  - St. Luke's Medical Center, Phoenix, Arizona
  - Memorial Medical Center, Modesto, California
  - Sutter Memorial Hospital, Sacramento, California
  - Christiana Care Health Services, Newark, Delaware
  - First Coast Cardiovascular Institute, P.A., Jacksonville, Florida
  - Augusta Vascular Center, Augusta, Georgia
  - DuPage Medical Group, Downers Grove, Illinois
  - Rockford Cardiovascular Associates, Rockford, Illinois
  - Central Iowa Hospital Corporation, Des Moines, Iowa
  - Cardiovascular Solutions, LLC, Shreveport, Louisiana
  - Sparrow Hospital, Lansing, Michigan
  - Mercy Hospital/Metropolitan Cardiology Consultants, Coon Rapids, Minnesota
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Wake Heart Research, Raleigh, North Carolina
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Lankenau Institute for Medical Research, Bryn Mawr, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - Sanford Research, Sioux Falls, South Dakota
  - Premier Surgical Associates, Knoxville, Tennessee
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Bellin Memorial Hospital, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Cohort: All patients enrolled in this study were treated with the EverFlex™ Self-Expanding Peripheral Stent System.
Period: Overall Study
Arm/Group | Study Cohort
Started | 108
Completed | 83
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | Study Cohort
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.06 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 88
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 108

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome - Freedom From Acute Death, Freedom From 36-month Amputation, and Freedom From 36-month Clinically-driven Target Lesion Revascularization
Description: Composite endpoint defined as freedom from acute death, freedom from 36-month amputation, and freedom from 36-month clinically-driven target lesion revascularization compared to a PTA performance goal.
Time Frame: 3 Years
Population: Subjects experiencing primary outcome within 3 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 108
Participants
  Subjects experiencing safety composite at 1 Year | 15
  Subjects experiencing safety composite at 2 Years | 23
  Subjects experiencing safety composite at 3 Years | 24
Statistical Analysis 1: Comparison: Study Cohort; Test type: Other — Freedom from primary safety composite event at 36 months compared to a performance goal of 35%; p < 0.001, Log Rank; Kaplan Meier = 0.771, 97.5% CI 1-sided [lower limit 0.678]

2. Secondary Outcome: Secondary Outcome - Freedom From Stent Fracture
Description: Determined by x-ray at 1, 2 and 3 years using the following classifications:
  Class 0 - No strut fractures Class I - Single tine fracture Class II - Multiple tine fractures Class III - Stent fracture(s) with preserved alignment of the components Class IV - Stent fracture(s) with mal-alignment of the components Class V - Stent fracture(s) in a trans-axial spiral configuration
  AND the following categories:
  Category A - Restenosis ≤ 50% at site of fracture Category B - Restenosis ≥ 50% at site of fracture Category C - Occlusion at site of fracture Category D - Unable to determine
Time Frame: 1, 2 and 3 years
Population: There were 103 stents evaluated by the Stent Fracture Adjudication Committee.
Measure: Number; unit: Stent
Arm/Group | Study Cohort
Number analyzed (Participants) | 103
Stent
  Stent Fracture at 1 Year | 0
  Stent Fracture at 2 Years | 1
  Stent Fracture at 3 Years | 3
Statistical Analysis 1: Comparison: Study Cohort; Stent Fracture at 1 Year; Test type: Other — No hypothesis Testing for this endpoint; Kaplan Meier = 1.0, Standard Error of Mean 0
Statistical Analysis 2: Comparison: Study Cohort; Stent Fracture at 2 Years; Test type: Other — No hypothesis testing was done for this endpoint; Kaplan Meier = 0.989, Standard Error of Mean 0.01
Statistical Analysis 3: Comparison: Study Cohort; Stent Fracture at 3 Years; Test type: Other — No hypothesis testing was done for this endpoint; Kaplan Meier = 0.965, Standard Error of Mean 0.02

3. Secondary Outcome: Secondary Outcome - Freedom From Acute Death, Freedom From Amputation and Freedom From Clinically-driven Target Lesion Revascularization at 1 and 2 Years
Description: Defined as the absence of all-cause mortality occurring within 30-days, absence of any major amputation within 12-/24- months and the absence of any clinically-driven repeat invasive procedure, including angioplasty, stenting, endarterectomy, bypass, or thrombolysis, performed to open or increase the lumen diameter inside or within 10 mm of the previously treated lesion due to the return of clinical symptoms within 12-/24- months of the procedure.
Time Frame: 1 and 2 years
Measure: Number; unit: participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 108
participants
  Subjects experiencing safety composite at 1 Year | 15
  Subjects experiencing safety composite at 2 Years | 23
Statistical Analysis 1: Comparison: Study Cohort; Freedom from acute death, freedom from amputation and freedom from clinically-driven target lesion revascularization at 1 year; Test type: Other — No hypothesis testing was done at this endpoint; Kaplan Meier = 0.86, Standard Error of Mean 0.034
Statistical Analysis 2: Comparison: Study Cohort; Freedom from acute death, freedom from amputation and freedom from clinically-driven target lesion revascularization at 2 years; Test type: Other — No hypothesis testing was done for this endpoint; Kaplan Meier = 0.782, Standard Error of Mean 0.04

4. Secondary Outcome: Secondary Outcome - Freedom From 36-month Amputation
Description: Defined as the absence of any major amputation (removal of the target limb or a part of the target limb above the metatarsal line) within 36 months of the procedure.
Time Frame: 3 Years
Measure: Number; unit: participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 108
participants
  Subjects with major amputation within 1 Year | 0
  Subjects with major amputation within 2 Years | 1
  Subjects with major amputation within 3 Years | 1
Statistical Analysis 1: Comparison: Study Cohort; Estimate from freedom from major amputation through 3 years; Test type: Other — No hypothesis testing was done for this endpoint; Kaplan Meier = 0.99, Standard Error of Mean 0.01

5. Secondary Outcome: Secondary Outcome - Freedom From 36-month Clinically-driven Target Lesion Revascularization
Description: Defined as the absence of any clinically-driven repeat invasive procedure, including angioplasty, stenting, endarterectomy, bypass, or thrombolysis, performed to open or increase the lumen diameter inside or within 10 mm of the previously treated lesion due to the return of clinical symptoms within 36 months of the procedure.
Time Frame: 3 Years
Measure: Number; unit: participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 108
participants
  Subjects experiencing CD-TLR within 1 Year | 15
  Subjects experiencing CD-TLR within 2 Years | 22
  Subjects experiencing CD-TLR within 3 Years | 23
Statistical Analysis 1: Comparison: Study Cohort; Freedom from clinically-driven TLR through 3 Years; Test type: Other; Kaplan Meier = 0.781, Standard Error of Mean 0.04

6. Secondary Outcome: Secondary Outcome - Number of Participants Free From Acute Death
Description: Defined as the absence of all-cause mortality occurring within 30 days of the procedure.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 108
Participants | 108

7. Secondary Outcome: Secondary Outcome - Number of Successfully Implanted Stents
Description: Defined as the ability to deploy the stent as intended at the treatment site.
Time Frame: At procedure
Measure: Count of Units; unit: Implanted Stents
Units Other Than Participants: Implanted Stents
Arm/Group | Study Cohort
Number analyzed (Participants) | 108
Number analyzed (Implanted Stents) | 118
Implanted Stents | 118

8. Secondary Outcome: Secondary Outcome - Number of Participants With Improvement in Rutherford Clinical Category at 1 Year
Description: Defined as an improvement in clinical status indicated by a decrease of one or more in Rutherford Clinical Category compared to baseline.
Time Frame: 1 Year
Population: There were 95 participants that were evaluated for the Rutherford Clinical Category at 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 95
Participants | 88

9. Secondary Outcome: Secondary Outcome - Number of Participants With Improvement in Ankle-Brachial Index at 1 Year
Description: Defined as an increase in the ankle-brachial index (ABI) compared to baseline in subjects with compressible arteries and baseline ABI < 0.9.
Time Frame: 1 Year
Population: There were 71 participants that were evaluated for the Ankle-Brachial Index at 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 71
Participants | 62

10. Secondary Outcome: Secondary Outcome - Change in Score of Walking Impairment Questionnaire at 1 Year
Description: Defined as an increase in Walking Impairment Questionnaire score in subjects who did not have iliac disease treated at the time of the index procedure compared to baseline
  Scale Range: Minimum score 0 to maximum score 100 Higher values represent better outcomes
Time Frame: 1 Year
Population: The total number of participants in the study was 108; number of participants analyzed depends on the questionnaires completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Cohort
Number analyzed (Participants) | 108
score on a scale
  Change from Baseline Score for pain aching cramp: number analyzed (Participants) | 83
  Change from Baseline Score for pain aching cramp | 30.42 (41.70)
  Change from Baseline Walking Distance Score: number analyzed (Participants) | 76
  Change from Baseline Walking Distance Score | 28.08 (39.37)
  Change from Baseline Walking Speed Score: number analyzed (Participants) | 76
  Change from Baseline Walking Speed Score | 21.77 (33.20)
  Change from Baseline Stair Climbing Score: number analyzed (Participants) | 75
  Change from Baseline Stair Climbing Score | 21.83 (36.05)

11. Secondary Outcome: Secondary Outcome - Number of Adverse Events
Description: Number of Adverse Events in the study through 3 Years.
Time Frame: 3 Years
Measure: Number; unit: Adverse Events
Arm/Group | Study Cohort
Number analyzed (Participants) | 108
Adverse Events | 206

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Study Cohort
All-Cause Mortality (participants affected / at risk) | 8/108
Serious Adverse Events (participants affected / at risk) | 66/108
Other Adverse Events (participants affected / at risk) | 0/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Cohort (N=108)
Stenosis (General disorders) | 21 (31)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Acute myocardial infarction (Cardiac disorders) | 6 (6)
Angina pectoris (Cardiac disorders) | 6 (8)
Arrhythmia (Cardiac disorders) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (6)
Cardiac failure congestive (Cardiac disorders) | 5 (6)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Ischemic colitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 4 (4)
Gangrene (General disorders) | 1 (1)
Necrosis (General disorders) | 1 (1)
Obstruction (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vascular stent thrombosis (General disorders) | 4 (4)
Cellulitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Genital candidiasis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (8)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Vascular access site infection (Infections and infestations) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (2)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Restenosis (Injury, poisoning and procedural complications) | 18 (19)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (2)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 3 (3)
Liver function test increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Amputation stump pain (Nervous system disorders) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac operation (Surgical and medical procedures) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (1)
Leg amputation (Surgical and medical procedures) | 1 (1)
Regional chemotherapy (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Artery dissection (Vascular disorders) | 5 (5)
Embolism (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 8 (9)
Ischaemic limb pain (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2)
Peripheral ischaemia (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT01680835/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT01680835/SAP_001.pdf